CLINICAL TRIAL: NCT03288376
Title: SNORE (Smartphone Analyses of Nocturnal Obstruction by Respiratory Evaluation) SOUNDS
Acronym: SNORESOUNDS
Status: Completed | Type: Observational
Sponsor: Incyphae, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SNORE_SOUNDS
Record Dates: First submitted 2017-09-13; First posted 2017-09-20 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Sleep Apnea, Obstructive; Chronic Obstructive Pulmonary Disease
Keywords: obstructive sleep apnea; polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective multipart clinical performance study to compare the ability of the SnoreSounds algorithm with polysomnography (PSG) and a type III Home Sleep Testing (HST) device to identify patients with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Consecutive patients referred to a sleep lab for possible OSA (obstructive sleep apnea) will be offered participation in this study. Study subjects will participate in either Part A, Part B or Part C of the study. Subjects will not participate in more than one part of the study. Study sites can participate in multiple parts of the study.

Part A: Sleep Lab

Consecutive patients referred to a sleep lab for possible OSA will be offered participation. Participants who provide informed consent will fill out a questionnaire and then have PSG, as it would normally be performed. During PSG additional sound recordings will be made in three ways:

1. Microphone placed 50-100 cm (20-40 inches) from the patient's mouth.
2. Android type Smart Phone with a recording application (app). The phone will be placed on a table 50-100 cm (20-40 inches)) from patient's mouth.
3. iPhone type Smart Phone with a recording app. Phone will be placed on a table 50-100 cm (20-40 inches) from patient's mouth.

The sound recordings obtained via the microphone and Smart Phones will be analyzed electronically for OSA by the sponsor's proprietary algorithm. A blinded comparison will be made between the PSG results and SnoreSounds algorithm results.

PSG will be performed and scored in a manner consistent with current (2012) American Academy of Sleep Medicine (AASM) standards. PSGs will be scored twice - with each scoring performed independently. If the Apnea Hypopnea Index (AHI) for each score places the patient in the same OSA severity range [0-4 normal/minimal OSA, 5-14 mild, 15-30 moderate, >30 severe] the average of the two scores will be utilized. If however the scores put the patent in different OSA severity ranges, then the study will be scored by an independent sleep medicine physician-sleep technician team and assigned an AHI.

The results of the SnoreSounds testing will not be known to the sleep lab and the results obtained from Snore Sounds analysis will not be utilized in the clinical management of study participants.

Part B: Comparison of SnoreSounds algorithm to Home Sleep Testing (HST) (currently not enrolling in Part B)

Part C: Comparison of SnoreSounds algorithm to Home Sleep Testing (HST) and to Polysomnography (PSG) (currently not enrolling in Part C)

ELIGIBILITY:
Inclusion Criteria:

* Patients >or= 18 years old who are referred for polysomnography (PSG) or Home Sleep Test (HST) because of possible obstructive sleep apnea (OSA)

Exclusion Criteria:

* Previous PSG or HST confirming OSA
* Prior surgery for snoring or OSA
* Medical contraindication for PSG
* Cognitive impairment that might interfere with obtaining informed consent or completing Clinical Questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women aged >or= 18 years who are referred for polysomnography (PSG) or Home Sleep Test (HST) because of possible obstructive sleep apnea (OSA).
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2015-02-13 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Agreement between algorithm with PSG reference standard for detection of OSA at an AHI cut-off of 15 | immediate
  Agreement between algorithm with PSG reference standard for detection of OSA at an AHI cut-off of 15

SECONDARY OUTCOMES:
Comparison between algorithm and PSG assignment of OSA severity based on AHI [0-4 normal/minimal OSA, 5-14 mild, 15-30 moderate, >30 severe]. | immediate
  Comparison between algorithm and PSG assignment of OSA severity based on AHI [0-4 normal/minimal OSA, 5-14 mild, 15-30 moderate, >30 severe].

CONTACTS AND LOCATIONS:
Overall Officials: Ruchir Sehra, MD, Principal Investigator — Incyphae, Inc.
Locations (3):
- United States (3):
  - Peninsula Sleep Center, Burlingame, California
  - Northeast Medical Group, New London, Connecticut
  - Doctors Community Hospital, Lanham, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pandian TNG, Sehra R, Narayan S. Breath variability increases in the minutes preceding obstructive sleep apneic events. Sleep Breath. 2021 Mar;25(1):271-280. doi: 10.1007/s11325-020-02094-1. Epub 2020 Jun 6. PMID 32506203
- [Derived] Narayan S, Shivdare P, Niranjan T, Williams K, Freudman J, Sehra R. Noncontact identification of sleep-disturbed breathing from smartphone-recorded sounds validated by polysomnography. Sleep Breath. 2019 Mar;23(1):269-279. doi: 10.1007/s11325-018-1695-6. Epub 2018 Jul 18. PMID 30022325